CLINICAL TRIAL: NCT05413226
Title: Effect of Different Ingestion Doses of Celastrol on Human Sperm Motility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legend Labz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AMT-001-2021
Record Dates: First submitted 2021-07-24; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Safety Issues
Keywords: sperm motility; sperm count; celastrol
MeSH Terms: interventions — celastrol

STUDY DESIGN:
Intervention Model Description: Healthy males from 18 to 40 years old
Masking Description: The participants will be masked to the dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amount of Celastrol Administered (Experimental): Increasing doses of Celastrol to each of five male subjects
  Interventions: Dietary Supplement: Celastrol

INTERVENTIONS:
Dietary Supplement: Celastrol — Four increasing doses of Celastrol to each of five men.
  Other Names: 24,25,26-trinoroleana-1(10),3,5,7- tetraen-29-oic acid

SUMMARY:
Five healthy participants with normal sperm counts and motility will ingest increasing doses of celastrol over a period of several days. After each dose ingestion the participants will provide an ejaculate the next day for sperm analysis. The objective is to see if increasing ingestion levels of celastrol will affect the sperm counts and motility of the participants.

DETAILED DESCRIPTION:
Experimental Design This will be an escalating dose study to determine the effects of different enteral dosages on sperm motility. Five healthy participants, of any ethnicity, between 18 and 40 years of age will be candidates for the study.

Baseline Days 1- 3 The five participants arrive at the clinic on Baseline Day 1, and will sign Consent Forms after being qualified by the inclusion and exclusion criteria. The participants will provide the first of three "qualifying" sperm samples (a sperm count of ~20 million sperm per milliliter of ejaculate, and sperm motility of ≥ 40% one hour after ejaculate). If the participants initial sample is "normal," then the participants will return to the clinic after three or more days to provide a second sperm sample. Again, if this second sample also meets the sperm count of ~20 million sperm per milliliter of ejaculate, and sperm motility of ≥ 40% one hour after ejaculate, then the participants will return to the clinic for a third time and provide a third and final "qualifying" sperm sample. The average of the "qualifying" sperm counts obtained during the three-day "qualifying period" will be used for the Baseline data, and will be used to compare sperm counts of the participants who ingest Celastrol during the remaining Experimental Days.

Experimental Day 1 All participants that provide three sperm samples that meet the "qualifying" criteria, will then return to the clinic after three or more days and have the participant medical histories taken; receive a physical examination; and have a blood sample taken. The five participants will be instructed to ingest the first dose of Celastrol (6.7 mg). Three hours after ingestion of this dose, the participants will provide a sperm sample.

Experimental Day 2 The participants will return to the clinic three days (or more) after Experimental Day 1. The five participants will be instructed to ingest the second dose of Celastrol (20.1 mg). Three hours after ingestion of this dose, the participants will provide another sperm sample.

Experimental Day 3 The participants will return to the clinic three days (or more) after Experimental Day 2. The five participants will be instructed to ingest the third dose of Celastrol (40.2 mg). Three hours after ingestion of this dose, the participants will provide another sperm sample.

Experimental Day 4 The participants will return to the clinic three days (or more) after Experimental Day 3. The five participants will be instructed to ingest the fourth dose of Celastrol (67.0 mg). Three hours after ingestion of this dose, the participants will provide another sperm sample.

The doses will be:

6.7 mg Commercial Dosage 20.1 mg 3x the Commercial Dose 40.2 mg 6x the Commercial Dose 67.0 mg 10x the Commercial Dose

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 40 years of age and who are found to be healthy without any underlying medical conditions that could affect sperm motility, and are not taking any daily medications. This does not exclude patients who take drugs prn.
2. Individuals who have not be involved in other clinical trials during the last 90 days. -

Exclusion Criteria:

1. Individuals who have been involved in any other clinical trial during the last 90 days.
2. Individuals who have sperm counts lower than that considered "normal." i.e. a sperm count of ~20 million sperm per milliliter of ejaculate, and (b) sperm motility of ≥ 40% one hour after ejaculate.
3. Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina
4. Individuals on medications that the clinician feels may affect sperm motility and/or otherwise interfere with the results
5. Medications that might interfere with blood chemistry, or CBCs
6. Subjects who are taking daily medications. The use of therapies prn is allowed.
7. Subjects Less than 18 years of age or over 40 years of age
8. Prisoners
9. Subjects who have taken anabolic steroid or testosterone during the last six months.
10. Subjects with a current history of addictive alcohol or illegal drug abuse (e.g. cocaine, heroin, etc.).

    The use of marijuana is allowed, but not preferred.
11. Subjects who are taking 5-alpha-reductase inhibitors (finasteride (Propecia®) and dutasteride (Avodart®), or Chemotherapy: -
12. Smokers

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-Smoking Healthy Males
Enrollment: 5 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Motility of Sperm in 1 mL of Ejaculate after Celastrol Ingestion | One Month
  Sperm samples will be analyzed independently for sperm motility
Amount of Sperm in 1 mL of Ejaculate after Celastrol Ingestion | One Month
  Sperm samples will be analyzed independently for number of sperm

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Patel, MD, Principal Investigator — Legend Labz, Inc.
Locations (1):
- Patient Urgent Care Clinic, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No